CLINICAL TRIAL: NCT00354380
Title: Safety and Efficacy of Methylene Blue Combined With Artesunate or Amodiaquine for Malaria Treatment in Children of Burkina Faso: a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFB544-A8-ASMB2006
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2006-10-24 (Estimated); Status verified 2006-09

CONDITIONS: Malaria
Keywords: Malaria; Africa; Methalyne-blue; Artesunate; Amodiaquine
MeSH Terms: conditions — Malaria | interventions — Methylene Blue; Artesunate; Amodiaquine

INTERVENTIONS:
Drug: Methylene blue
Drug: Artesunate
Drug: Amodiaquine

SUMMARY:
The primary objective of this trial is to study the safety of the combination methylene blue (MB)-artesunate (AS) and MB-amodiaquine (AQ) in treating malaria among children compared to the safety of an AS-AQ regimen. The secondary objective is to investigate the efficacy of MB-AS and MB-AQ.

DETAILED DESCRIPTION:
Objectives: The primary objective of this trial is to study the safety of the combination methylene blue (MB)-artesunate (AS) and MB-amodiaquine (AQ) given over three days in 6-10 year old children with uncomplicated falciparum malaria in a malaria endemic area compared to the safety of a three days AS-AQ regimen. Secondary objectives are to investigate the efficacy of MB-AS and MB-AQ.

Population: Children aged 6-10 years with uncomplicated malaria from Nouna town.

Sample size: N= 180 (n=60 for each group).

Treatment: The participants in the MB-AS group will receive orally twice daily 9mg/kg MB combined with once daily 4mg/kg AS over 3 days. The participants in the MB-AQ group will receive orally twice daily 9mg/kg MB combined with once daily 10mg/kg AQ over 3 days. The participants of the comparator group will receive a 3 day regimen of once daily oral AS (4mg/kg) combined with once daily AQ (10mg/kg).

Endpoints: The primary endpoint is the number of adverse events (AE) after drug intake until day 28. Secondary endpoints are the number of serious adverse events (SAE), adequate clinical and parasitological response (ACPR) rate on day 28, clinical and parasitological failure rates on day 3, 7, 14 and 28, changes in haematocrit until day 28, and fever and parasite clearance time.

ELIGIBILITY:
Inclusion criteria:

* 6-10 year old children
* Ability to swallow tablets
* Uncomplicated malaria caused by P. falciparum
* Asexual parasites ≥ 2000/µl and < 200000/µl
* Axillary temperature ≥ 37.5°C
* Burkinabe nationality
* Informed consent

Exclusion Criteria:

* Complicated or severe malaria
* Any apparent significant disease
* Anaemia (haematocrit < 21%)
* Treated in the same trial before
* Antimalarial treatment prior to inclusion (last three days), except children having been treated with chloroquine

Ages: 6 Years to 10 Years | Sex: All
Age Groups: Child
Dates: Start 2006-09; Study Completion 2006-11

PRIMARY OUTCOMES:
Incidence of observed and self-reported non-serious adverse events over the 28 days observation period (definition chapter 11)

SECONDARY OUTCOMES:
Incidence of serious adverse events (definition: chapter 11) over the 28 days observation period
ACPR rate until D28
Early treatment failure (ETF) rate
Late clinical failure (LCF) rate at D14 and D28
Late parasitological failure (LPF) rate at D14 and D28
Fever clearance time
Parasite clearance time
Change in haematocrit after 2, 3, 7, 14 and 28 days compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Mueller, MD, MPH, Principal Investigator — Heidelberg University; Peter Meissner, MD, MSc Trop Paed, Principal Investigator — Heidelberg University
Locations (1):
- Nouna District Hospital, Nouna, Burkina Faso

REFERENCES:
- [Derived] Coulibaly B, Zoungrana A, Mockenhaupt FP, Schirmer RH, Klose C, Mansmann U, Meissner PE, Muller O. Strong gametocytocidal effect of methylene blue-based combination therapy against falciparum malaria: a randomised controlled trial. PLoS One. 2009;4(5):e5318. doi: 10.1371/journal.pone.0005318. Epub 2009 May 5. PMID 19415120
- [Derived] Zoungrana A, Coulibaly B, Sie A, Walter-Sack I, Mockenhaupt FP, Kouyate B, Schirmer RH, Klose C, Mansmann U, Meissner P, Muller O. Safety and efficacy of methylene blue combined with artesunate or amodiaquine for uncomplicated falciparum malaria: a randomized controlled trial from Burkina Faso. PLoS One. 2008 Feb 20;3(2):e1630. doi: 10.1371/journal.pone.0001630. PMID 18286187